CLINICAL TRIAL: NCT03166098
Title: The Role of Dysmyelination in Cognitive Impairment of Psychotic Spectrum Disorders
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 15-00754
Record Dates: First submitted 2017-05-23; First posted 2017-05-24 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Schizophrenia; Bipolar Disorder
Keywords: Psychotic Spectrum Disorders
MeSH Terms: conditions — Schizophrenia; Bipolar Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Diagnosis of Schizophrenia
  Interventions: Diagnostic Test: Cognitive Function Assessments
- Diagnosis of Bipolar Disorder
  Interventions: Diagnostic Test: Cognitive Function Assessments
- Unaffected siblings of the SZ groups
  Interventions: Diagnostic Test: Cognitive Function Assessments
- Unaffected siblings of the BP group
  Interventions: Diagnostic Test: Cognitive Function Assessments
- Healthy control (HC) comparison group
  Interventions: Diagnostic Test: Cognitive Function Assessments

INTERVENTIONS:
Diagnostic Test: Cognitive Function Assessments — The NIMH-Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) is a consensus battery that is considered state-of-the art in the evaluation of cognitive skills for schizophrenia research.(Burton et al., 2013, Harvey, 2014) The complete cognitive battery takes about one hour to administer, and is comprised of 10 subtests measuring seven essential domains of function, with very good reliability and validity.(Nuechterlein 2008, August et al., 2012) The MATRICS subtests have been incorporated into the cognitive battery described below, with supplementary subtests included where indicated within each domain.

SUMMARY:
This is a single center study that uses both between-group comparisons and correlational analyses to establish biomarkers of dysmyelination and cognitive impairment in Psychotic Spectrum Disorders using imaging and neuropsychological assays.The study will provide non-invasive biomarkers of cognitive dysfunction in Psychotic Spectrum Disorder.

ELIGIBILITY:
Inclusion Criteria:

Patients:

* current DSM-5-defined diagnosis of a schizophrenia or bipolar disorder. A best estimate diagnostic approach will be utilized in which information from the Diagnostic Interview for Genetic Studies (DIGS) is supplemented by information from family informants, psychiatrists, and medical records to generate a diagnosis as needed
* no alcohol or substance abuse during the last 6 month
* no current substance-induced psychotic disorder or a psychotic disorder due to a general medical condition determined by DSM-5 criteria
* ages 18 to 30 years old;
* any race
* competent and willing to sign informed consent
* within 5 years from the disease onset.

Siblings:

* have the same biological parents as their PSD sibling
* any race
* no current or past history of psychotropic medication usage
* no alcohol or substance abuse during the last 6 months
* competent and willing to sign informed consent;
* ages 18 to 30 years old.

Healthy controls:

* matched for age to PSD patients
* no current or past history of psychotropic medication usage
* no prodromal symptoms and no family history of PSD
* no alcohol or substance abuse during the last 6 months
* competent and willing to sign informed consent.
* all attempts will be made to recruit controls with similar parental SES as patients. However, given that PSD are both a neurodevelopmental and familial disorder, exact matching for educational level or IQ may neither be possible nor desirable.

have the same biological parents as their PSD sibling

* any race
* no current or past history of psychotropic medication usage
* no alcohol or substance abuse during the last 6 months
* competent and willing to sign informed consent;
* ages 18 to 30 years old.

Exclusion Criteria:

* a serious neurological or endocrine disorder or any medical condition or treatment known to affect the brain, 2) organic brain disorder, mental retardation, or significant medical illness;
* significant risk of suicidal or homicidal behavior;
* must not have met DSM-5 criteria for current alcohol or drug dependence in the last 6 months;
* contraindications to MRI scanning (i.e., metal implants, pacemakers, pregnancy, etc.);
* documented loss of consciousness (LOC) for longer than 30 minutes or LOC with any neurological sequelae.

Ages: 18 Years to 30 Years | Sex: All
Age Groups: Adult
Study Population: The study will include patients with a diagnosis of Schizophrenia or Bipolar Disorder with Psychotic features, their unaffected siblings, and comparison healthy subjects.
Sampling Method: Non-Probability Sample
Enrollment: 139 (Actual)
Dates: Start 2016-07-05 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
DKI(metrics RDextra, faxon, and ADextra) Metrics | 6 Years
  To compare DKI metrics (faxon, RDextra, and ADextra) in patients with SZ or BP, their unaffected siblings (SIB), and healthy comparison control (HC) subjects
Magnetic Resonance Spectroscopy will be employed to obtain quantitative metrics of choline (Cho) | 1 Hour
  Choline Concentration (1H-MRS)

CONTACTS AND LOCATIONS:
Overall Officials: Mariana Lazar, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States